CLINICAL TRIAL: NCT02314377
Title: Bevacizumab Therapy for Brain Arteriovenous Malformation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Daniel L. Cooke, Associate Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNA1052
Record Dates: First submitted 2014-11-25; First posted 2014-12-11 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Brain Arteriovenous Malformation
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AVM treatment with Bevacizumab (Experimental): Bevacizumab infusion dose of 5mg/kg q 2 weeks for 12 weeks (2.5 mg/week).
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab dosing of 5mg/kg q 2 weeks for 12 weeks (2.5 mg/week).
  Other Names: avastin

SUMMARY:
Bevacizumab Therapy for brain arteriovenous malformation that is not amenable to surgical intervention.

DETAILED DESCRIPTION:
Brain AVMs are relatively rare, though their potential for ICH along with the existence of effective treatments makes their diagnosis and management essential to the community. The 2-4% annual incidence of such secondary ICH creates controversy regarding treatment for asymptomatic patients. Brain AVMs thus require multidisciplinary evaluation for optimal management especially for surgical grades III - V lesions that often require some combination of embolization, microsurgery, and/or radiosurgical treatment. Currently there is no designated medical therapy for bAVM, though there is growing animal and human evidence supporting a role for bevacizumab to reduce the size of AVMs in the brain and liver, respectively. This proposal is a pilot study to assess the efficacy and safety of bevacizumab in humans with bAVMs.

ELIGIBILITY:
Inclusion Criteria:

* bAVM deemed unsuitable for invasive treatment OR patient has elected to defer invasive treatment OR failed conventional therapy
* Age greater than 18 years at time of first study drug administration
* Spetzler-Martin grade III - V
* Progressive or disabling signs and symptoms as determined by the study investigators. In the case of sporadic bAVM, these would be referable to the lesion, e.g., progressive neurological deficits, refractory headaches and seizures; for HHT patients, bAVM may be asymptomatic, but patient must have one progressively symptomatic manifestation of HHT that is referable to a vascular lesion, e.g., epistaxis, GI bleeding; or another solid organ AVM
* Patients must have adequate bone marrow function (WBC > 3,000/μl, ANC > 1,500/mm3, platelet count of > 100,000/mm3, and hemoglobin > 10 mg/dl), adequate liver function (SGOT and bilirubin < 1.5 times ULN), and adequate renal function (creatinine < 1.5 mg/dL) within 14 days before starting therapy
* Negative pregnancy test within 14 days of starting therapy
* Patients must not have proteinuria at screening as demonstrated by either 1) urine protein: creatinine (UPC) ratio > 1.0 at screening, OR 2) urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible)
* Patients must not have inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg) on antihypertensive medications
* Patients must not have any prior history of hypertensive crisis or hypertensive encephalopathy
* Patients must not have New York Heart Association Grade II or greater congestive heart failure
* Patients must not have history of myocardial infarction or unstable angina within 12 months prior to study enrollment
* Patients must not have symptomatic peripheral vascular disease
* Patients must not have significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Patients must not have major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks of beginning Avastin or the anticipation of need for major surgical procedure during the course of the study
* Patients must not have core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to bevacizumab
* Patients must not have a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Patients must not have serious, non-healing wound, ulcer, or bone fracture
* Patients must not be pregnant or breast-feeding. Women of childbearing potential are required to obtain a negative pregnancy test within 14 days of starting treatment. Effective contraception (men and women) must be used in subjects of child-bearing potential
* Patients must not be on any other experimental agents/clinical trials
* Signed informed consent

Exclusion Criteria:

* Diffuse lesion that cannot be assessed in terms of volume by cross-sectional imaging on MRI
* Inability to undergo MRI scans
* Coagulation disorders, e.g., thrombocytopenia, coagulopathy or anticoagulant therapy (Plavix and ASA is not excluded)
* Low probability to adhere to study protocol or functional impairment that could compromise safety monitoring
* Unstable medical or psychiatric illness
* Ovarian dysfunction (criteria waived if potential future to have children (e.g. post menopausal or s/p tubal ligation) limited biologically.
* Clinically significant thrombotic episode within the last 24 weeks
* Atrial fibrillation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06; Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Our primary outcome will be change in AVM volume from pre-treatment MRI. | 12, 26 and 52 weeks
  AVM volume will be assessed by review of standardized 1.5 mm slices in the axial plane. The contour of the vascular mass using time-of-flight MR angiography sequences will generate a cross-sectional area at each slice level. The volume will be estimated by summing the imputed volume of each slice. This is the standard method in radiation oncology used to assess bAVM volume for radiosurgery treatment planning using commercial software (Leksell GammaPlan). The source images and measurement images will be archived on a research workstation. After a baseline MR examination, follow-up MRs will be performed at 12, 26 and 52 weeks.

SECONDARY OUTCOMES:
Serum VEGF levels | at baseline and at 12, 26 and 52 weeks
Urine analysis | at baseline and at 12, 26 and 52 weeks
Physical exam | at baseline and at 12, 26 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cooke, MD, Principal Investigator — UCSF Medical Center
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Muster R, Ko N, Smith W, Su H, Dickey MA, Nelson J, McCulloch CE, Sneed PK, Clarke JL, Saloner DA, Eisenmenger L, Kim H, Cooke DL. Proof-of-concept single-arm trial of bevacizumab therapy for brain arteriovenous malformation. BMJ Neurol Open. 2021 Mar 17;3(1):e000114. doi: 10.1136/bmjno-2020-000114. eCollection 2021. PMID 34189463